CLINICAL TRIAL: NCT04312282
Title: An Open-Label Study of the Effect of Tesetaxel on the QTc Interval and the Effect of Food, Itraconazole, and Rifampin on Tesetaxel Pharmacokinetics in Patients With Advanced Solid Tumors
Brief Title: The Effect of Tesetaxel on the QTc Interval and the Effect of Food, Itraconazole, and Rifampin on Tesetaxel Pharmacokinetics in Patients With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The Sponsor has discontinued the development of tesetaxel
Sponsor: Odonate Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ODO-TE-S101
Record Dates: First submitted 2020-03-13; First posted 2020-03-18 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Advanced Solid Tumors
Keywords: tesetaxel; itraconazole; rifampin; food effect; QTc interval; food-drug interaction; drug-drug interaction; PK; tesetaxel metabolites; advanced solid tumor
MeSH Terms: interventions — tesetaxel; Itraconazole; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1, Sequence 1A: Fed then fasted (Experimental): Cycle 1: Tesetaxel on Day 1 of a 21-day cycle under fed conditions
  Cycle 2: Tesetaxel on Day 1 of a 21-day cycle under fasted conditions
  Interventions: Drug: Tesetaxel
- Cohort 1, Sequence 1B: Fasted then fed (Experimental): Cycle 1: Tesetaxel on Day 1 of a 21-day cycle under fasted conditions
  Cycle 2: Tesetaxel on Day 1 of a 21-day cycle under fed conditions
  Interventions: Drug: Tesetaxel
- Cohort 2: Tesetaxel plus itraconazole (Experimental): Cycle 1: Tesetaxel on Day 1 of a 21-day cycle
  Cycle 2: Tesetaxel on Day 1 of a 21-day cycle and itraconazole on Day -3 through Day 14 of a 21-day cycle
  Interventions: Drug: Tesetaxel; Drug: Itraconazole
- Cohort 3: Tesetaxel plus rifampin (Experimental): Cycle 1: Tesetaxel on Day 1 of a 21-day cycle
  Cycle 2: Tesetaxel on Day 1 of a 21-day cycle and rifampin on Day -6 through Day 14 of a 21-day cycle
  Interventions: Drug: Tesetaxel; Drug: Rifampin

INTERVENTIONS:
Drug: Tesetaxel — Tesetaxel orally on Day 1 of a 21-day cycle
  Arms: Cohort 1, Sequence 1A: Fed then fasted
Drug: Tesetaxel — Tesetaxel orally on Day 1 of a 21-day cycle
  Arms: Cohort 1, Sequence 1B: Fasted then fed; Cohort 2: Tesetaxel plus itraconazole; Cohort 3: Tesetaxel plus rifampin
Drug: Itraconazole — Itraconazole orally once daily from Day -3 to Day 14 of a 21-day cycle
  Arms: Cohort 2: Tesetaxel plus itraconazole
Drug: Rifampin — Rifampin orally once daily from Day -6 to Day 14 of a 21-day cycle
  Arms: Cohort 3: Tesetaxel plus rifampin

SUMMARY:
This is a 3-cohort, multicenter, Phase 1 study of the effect of tesetaxel, an investigational, orally administered taxane, on the corrected QT (QTc) interval and the potential effect of food, a cytochrome P450 (CYP) 3A inhibitor (itraconazole), and a CYP3A inducer (rifampin) on tesetaxel pharmacokinetics (PK) in adult patients with advanced solid tumors.

DETAILED DESCRIPTION:
Cohort 1:

Cohort 1 is a 2-period, 2-sequence, crossover study designed to assess the effect of food on the PK of tesetaxel and tesetaxel metabolites. Patients were randomized in a 1:2 ratio to receive tesetaxel on Day 1 of two 21-day cycles under fed and fasting conditions in one of two opposing sequences (Sequence 1A and Sequence 1B).

Cohort 2:

Cohort 2 is a 2-period, single-sequence, crossover study designed to assess the potential PK drug-drug interaction (DDI) of a strong CYP3A inhibitor (itraconazole) on tesetaxel and tesetaxel metabolites. Patients receive tesetaxel during Cycle 1 followed by a reduced dose of tesetaxel plus itraconazole during Cycle 2.

Cohort 3:

Cohort 3 is a 2-period, single-sequence, crossover study designed to assess the potential PK DDI of a strong CYP3A inducer (rifampin) on tesetaxel and tesetaxel metabolites. Patients receive tesetaxel during Cycle 1 followed by tesetaxel plus rifampin during Cycle 2.

Patients in all cohorts also participate in a study designed to assess the effect of tesetaxel and tesetaxel metabolites on cardiac repolarization as measured by the change from baseline in the QTc interval over the first cycle of treatment. Patients who are tolerating and benefitting from treatment with tesetaxel have the opportunity to continue onto an optional treatment extension.

ELIGIBILITY:
Inclusion Criteria:

* Female or male patients at least 18 years of age
* Histologically or cytologically confirmed solid tumor
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1 or 2
* Adequate cardiac conduction by ECG
* Adequate bone marrow, hepatic, and renal function

Exclusion Criteria:

* Presence of risk factors for QTc prolongation
* Presence of neuropathy Grade > 1
* Anticancer treatment ≤ 14 days prior to randomization
* Major surgery ≤ 28 days prior to randomization
* Less than 2 weeks or 5 plasma half-lives (whichever is greater) since last use of:

  * A moderate or strong inhibitor or inducer of CYP3A
  * A CYP3A substrate with a narrow therapeutic range or that is contraindicated with either itraconazole or rifampin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2020-03-06 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
All Cohorts: The change from baseline in Fridericia's corrected QT (ΔQTcF) interval | Approximately 3 weeks
Cohort 1, Sequences 1A and 1B: Maximum observed plasma concentration (Cmax) for tesetaxel under fed and fasted conditions | Approximately 6 weeks
Cohort 1, Sequences 1A and 1B: Area under the plasma concentration-time curve from 0 to the last measurable plasma concentration (AUC0-t) for tesetaxel under fed and fasted conditions | Approximately 6 weeks
Cohort 2: Cmax for tesetaxel in the presence and absence of itraconazole | Approximately 6 weeks
Cohort 2: AUC from 0 to 336 hours (AUC0-336h) for tesetaxel in the presence and absence of itraconazole | Approximately 6 weeks
Cohort 3: Cmax for tesetaxel in the presence and absence of rifampin | Approximately 6 weeks
Cohort 3: AUC0-336h for tesetaxel in the presence and absence of rifampin | Approximately 6 weeks

SECONDARY OUTCOMES:
All Cohorts: Cmax for tesetaxel metabolites | Approximately 6 weeks
All Cohorts: AUC for tesetaxel metabolites | Approximately 6 weeks
All Cohorts: Treatment-emergent adverse events (TEAEs), including serious adverse events (SAEs) | Baseline through 30 days after last administration of Study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Joseph O'Connell, M.D., Study Director — Odonate Therapeutics, Inc.
Locations (3):
- United States (3):
  - START Midwest, Grand Rapids, Michigan
  - Mary Crowley Cancer Research, Dallas, Texas
  - NEXT Oncology, San Antonio, Texas